CLINICAL TRIAL: NCT05616065
Title: Bias Reduction in Academic Recruitment
Acronym: BRIAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Community Medical Center, Toms River, NJ (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-029
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Internship and Residency; Interview; Education, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blinded (Experimental): Interviewers will be assigned a candidate to interview. They will be asked not to review the medical school transcripts or standardized test scores (USMLE, COMLEX). They will be permitted to review personal statements, letters or recommendation, and other personal information in the application.
  Interventions: Other: Blinding to academic performance of candidate
- Unblinded (Active Comparator): Interviewers will be assigned a candidate to interview. They will be given full permission to review the full application of their candidate as per their normal interview protocol.
  Interventions: Other: Usual Interview methodology

INTERVENTIONS:
Other: Blinding to academic performance of candidate — Each candidate applying to our program will be interviewed by three core faculty. One of them will be selected, a priori, to be asked not to view a candidate's academic performance (medical school transcripts, standardized test scores). This will not be randomized. Instead, it shall be set up so that each assessor has two blinded candidates to interview each day scheduled. Given that different faculty will be scheduled each day, it may end up that certain faculty will be blinded more than others.
  Arms: Blinded
Other: Usual Interview methodology — Each candidate applying to our program will be interviewed by three core faculty. Two of them will be selected, a priori, to be asked to interview their candidates as they see fit.
  Arms: Unblinded

SUMMARY:
The aim of this study is to determine if, with respect to medical students applying for residency in emergency medicine, prior knowledge of an applicant's academic record affects their ranking during their interviews.

Attendings interviewing candidates will either be blinded to their prior academic records or be allowed to review them prior to the interview. The interviewer's final score of the applicant will be measured, comparing blinded versus unblinded assessors.

DETAILED DESCRIPTION:
In residency recruitment and ranking, the most honest admission educators can offer is that there truly is no exact way to identify candidates who will thrive in a given discipline or residency program. Along with applications and letters of reference, the traditional residency interview process has long been thought to be one of the best available tools to evaluate a given candidate as well as assess their 'fit' for the culture of the program they wish to enter. Despite this decades-used tool, little uniformity exists in practice, with various disciplines and programs using various techniques to evaluate potential residents. To wit, prospective resident themselves, in one study, have listed their top three consideration when selecting a residency to be the friendliness of the program and faculty, the overall environment, and the interview day itself. Spending time in the department and hospital and having contact with the faculty and staff has long been seen as the best way to 'get to know' the program. This is among the main reasons why medical students will often schedule 'audition rotations' at hospitals and programs that draw their interest.

With respect to the interviews themselves, there has been some evolution of thought, despite the variability. Recently, structured interviews and other techniques have been discussed to reduce bias and increase efficiency in residency recruitment.

While this has been discussed in academic circles for some time, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has brought these issues to the fore. Forcing interviews to be done remotely has effectively removed the intimacy of an in-person visit or interview, making an assessment of 'fit' for both the applicant and the program more challenging. Many program leaders and resident educators have described 'fit' as among the most important predictors of residency success, sometimes more so than pure academic prowess.

Of the many biases in residency interviewing, among the easiest and most seductive is hinging a decision on academic achievement alone. It is well understood by many residency educators that academic success in medical school does not always translate to the same level of performance in residency. With the virtual method of interviews continuing for at least this year (and likely going forward), our study ponders the question if the removal of knowledge of an applicant's academic record changes their interviewer's perception of their potential as a resident in an emergency medicine.

This study will examine if blinding interviewers to the academic performance of residency applicants impact the assessor's recommendation for the candidate's match day rank list placement. Candidates will be assigned to have one of three of their interviews performed during the standard interview process, to have a single assessor who is instructed not to look at either medical school transcripts or standardized test scores. Assessors will be permitted to look at letters of recommendation, personal statements, research and work experience, and hobbies.

The absolute value of the difference of between blinded and unblinded assessors will be compared and tested for statistical significance by matched student T testing. The study is powered for an absolute difference of 1 point on a ten-point scale, which translates linearly to rank list placement. Additionally, this 1-point difference is considered significant from a standpoint of residency operations. Also, blinded versus unblinded assessors will be compared to the placement by the residency program director, who will remain unblinded and also makes independent recommendations for every candidate. As a subanalysis, a qualitative assessment of candidates who get ranked either substantially higher or lower when blinded compared to unblinded will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* All candidates who have or are anticipating completing their medical school education, and have applied for a position in our residency during the 2022-2023 match cycle.

Exclusion Criteria:

* Candidates our program declined to grant an interview spot or have canceled their interview prior to completing it.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Assessor recommendation for match list position | Immediately after interview
  Assessors will be asked to score their applicant, 1-10, with 1 corresponding to a Do Not Rank recommendation, 2-4 with lower third of list, 5-7 middle third of list, and 8-10 upper third of list.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Kravitz, MD, Principal Investigator — Associate Program Director, Emergency Medicine Residency
Locations (1):
- Community Medical Center, Toms River, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiraly L, Dewey E, Brasel K. Hawks and Doves: Adjusting for Bias in Residency Interview Scoring. J Surg Educ. 2020 Nov-Dec;77(6):e132-e137. doi: 10.1016/j.jsurg.2020.08.013. Epub 2020 Aug 27. PMID 32863174
- [Background] Poon S, Nellans K, Rothman A, Crabb RAL, Wendolowski SF, Kiridly D, Gecelter R, Gorroochurn P, Chahine NO. Underrepresented Minority Applicants Are Competitive for Orthopaedic Surgery Residency Programs, but Enter Residency at Lower Rates. J Am Acad Orthop Surg. 2019 Nov 1;27(21):e957-e968. doi: 10.5435/JAAOS-D-17-00811. PMID 30614894
- [Background] Hughes RH, Kleinschmidt S, Sheng AY. Using structured interviews to reduce bias in emergency medicine residency recruitment: Worth a second look. AEM Educ Train. 2021 Sep 1;5(Suppl 1):S130-S134. doi: 10.1002/aet2.10562. eCollection 2021 Sep. No abstract available. PMID 34616987
- [Background] Williams AL, Blomkalns AL, Gibler WB. Residency training in emergency medicine: the challenges of the 21st century. Keio J Med. 2004 Dec;53(4):203-9. doi: 10.2302/kjm.53.203. PMID 15647626
- [Background] Balhara KS, Weygandt PL, Ehmann MR, Regan L. Navigating Bias on Interview Day: Strategies for Charting an Inclusive and Equitable Course. J Grad Med Educ. 2021 Aug;13(4):466-470. doi: 10.4300/JGME-D-21-00001.1. Epub 2021 Aug 13. No abstract available. PMID 34434507
- [Background] Theiss LM, Prather JC, Porterfield JR, Corey B, Chen H, McGwin G, Johnson MD, Theiss SM. Prevalence, Bias, and Rank List Impact of Illegal Questions in Surgical Specialty Residency Interviews. J Surg Educ. 2022 Jan-Feb;79(1):69-76. doi: 10.1016/j.jsurg.2021.07.015. Epub 2021 Aug 13. PMID 34400121
- [Background] DeSantis M, Marco CA. Emergency medicine residency selection: factors influencing candidate decisions. Acad Emerg Med. 2005 Jun;12(6):559-61. doi: 10.1197/j.aem.2005.01.006. PMID 15930408
- [Background] Smilen SW, Funai EF, Bianco AT. Residency selection: should interviewers be given applicants' board scores? Am J Obstet Gynecol. 2001 Feb;184(3):508-13. doi: 10.1067/mob.2001.109868. PMID 11228511
- [Background] Haas MRC, He S, Sternberg K, Jordan J, Deiorio NM, Chan TM, Yarris LM. Reimagining Residency Selection: Part 1-A Practical Guide to Recruitment in the Post-COVID-19 Era. J Grad Med Educ. 2020 Oct;12(5):539-544. doi: 10.4300/JGME-D-20-00907.1. No abstract available. PMID 33149819
- [Background] Sternberg K, Jordan J, Haas MRC, He S, Deiorio NM, Yarris LM, Chan TM. Reimagining Residency Selection: Part 2-A Practical Guide to Interviewing in the Post-COVID-19 Era. J Grad Med Educ. 2020 Oct;12(5):545-549. doi: 10.4300/JGME-D-20-00911.1. No abstract available. PMID 33149820
- [Background] Jordan J, Sternberg K, Haas MRC, He S, Yarris LM, Chan TM, Deiorio NM. Reimagining Residency Selection: Part 3-A Practical Guide to Ranking Applicants in the Post-COVID-19 Era. J Grad Med Educ. 2020 Dec;12(6):666-670. doi: 10.4300/JGME-D-20-01087.1. Epub 2020 Dec 18. No abstract available. PMID 33391587
- [Background] Stephenson-Famy A, Houmard BS, Oberoi S, Manyak A, Chiang S, Kim S. Use of the Interview in Resident Candidate Selection: A Review of the Literature. J Grad Med Educ. 2015 Dec;7(4):539-48. doi: 10.4300/JGME-D-14-00236.1. PMID 26692964